CLINICAL TRIAL: NCT05555407
Title: A Pilot Study to Assess the Feasibility of a Wireless Patch System (WPS) to Measure Gastrointestinal Motility and Gastric Emptying
Brief Title: Feasibility of a Wireless Patch System (WPS) to Measure Gastrointestinal Motility and Gastric Emptying
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brian Lacy, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-004957
Record Dates: First submitted 2022-09-19; First posted 2022-09-26 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Gastric Emptying
Keywords: Scintigraphy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wireless patch system (WPS) (Experimental): Subjects scheduled for a gastric emptying scan will have a wireless patch system (WPS) placed.
  Interventions: Diagnostic Test: Scintigraphic gastric emptying scan; Device: Wireless patch system (WPS)

INTERVENTIONS:
Diagnostic Test: Scintigraphic gastric emptying scan — Nuclear medicine scan that provides an assessment of gastric motility
Device: Wireless patch system (WPS) — Wireless wearable patches applied to the abdomen after 3 small areas of the abdomen that connect to a recording device for a total of 6 days and subjects will track mealtimes, bowel movements, and sleep using an iPhone app.

SUMMARY:
The purpose of this study is to evaluate the utility of a new device - an external wireless patch system (WPS) - to measure gastric motility and to compare this external wearable device with the most commonly used test to measure stomach emptying, the nuclear medicine gastric emptying scan (also called gastric scintigraphy).

ELIGIBILITY:
Inclusion Criteria:

* Referred to the nuclear medicine department for a scintigraphic gastric emptying scan.

Exclusion Criteria:

* Have had prior gastric or esophageal surgery.
* Have had surgery to the GI tract within the last 60 days (e.g., appendectomy, cholecystectomy).
* Are on chronic opioids or other medications known to affect gastric emptying (e.g., GLP-1 agonists, high dose tricyclic agents).
* Have been recently hospitalized for complications of diabetes or have a HgbA1c > 10.
* Have severe psychological distress preventing study participation.
* Unable to read or understand the consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Subject willingness to wear a wireless patch system (WPS) | 7 days
  Number of subjects to wear a wireless patch system (WPS) to evaluate upper gastrointestinal symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Brian Lacy, PhD, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials